CLINICAL TRIAL: NCT00004045
Title: A Phase II Study of Intravenous DX-8951f Administered Daily for Five Days Every Three Weeks to Patients With Hormone-Refractory Prostate Cancer
Brief Title: Chemotherapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067146; DAIICHI-8951A-PRT012; SACI-IDD-99-03; SLLH-BHS-99-0020
Record Dates: First submitted 1999-12-10; First posted 2004-04-15 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Prostate Cancer
Keywords: stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — exatecan

INTERVENTIONS:
Drug: exatecan mesylate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of DX-8951f in treating patients who have metastatic prostate cancer that has not responded to hormone therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the antitumor activity of DX-8951f as measured by PSA response in patients with hormone refractory prostate cancer. II. Determine the antitumor activity of this drug in the subpopulation of these patients with measurable disease. III. Evaluate the quantitative and qualitative toxicities of this drug in these patients. IV. Evaluate the pharmacokinetics of this drug in these patients.

OUTLINE: This is a multicenter study. Patients receive DX-8951f IV over 30 minutes daily for 5 days. Courses repeat every 21 days. Treatment continues in the absence of unacceptable toxicity or disease progression. Patients with no evidence of PSA decrease by the start of course 3 receive no further treatment. Patients are followed every 3 months until death.

PROJECTED ACCRUAL: A total of 12-37 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed prostate carcinoma Metastatic disease Documented progression of prostate cancer while receiving androgen ablative therapy (i.e., surgical or chemical castration and a serum testosterone level in the castrate range) Documented hormone therapy resistance defined as: PSA rise on 3 occasions not less than 4 weeks apart Any evidence of progressive measurable disease PSA must be above 20 ng/mL prior to study entry No brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Hemoglobin at least 9.0 g/dL Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT/SGPT no greater than 2 times upper limit of normal (ULN) (5 times ULN if liver metastases present) Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No active congestive heart failure No uncontrolled angina No myocardial infarction within the past 6 months Other: Fertile patients must use effective contraception No uncontrolled pain requiring irradiation No concurrent serious infection No other malignancy within the past 5 years except nonmelanoma skin cancer No overt psychosis, mental disability, or incompetence

PRIOR CONCURRENT THERAPY: Biologic therapy: No prophylactic colony stimulating factors to prevent neutropenia No concurrent biologic therapy Chemotherapy: No more than 1 prior cytotoxic chemotherapy regimen No concurrent cytotoxic chemotherapy Endocrine therapy: See Disease Characteristics At least 6 weeks since prior peripheral antiandrogens (e.g., flutamide) No concurrent steroid therapy initiated within past 2 months Current LHRH agonist therapy should continue through study Radiotherapy: At least 4 weeks since prior radiotherapy (except low dose, non myelosuppressive) and recovered No prior irradiation to greater than 25% of bone marrow No prior strontium chloride Sr 89 or samarium Sm 153 lexidronam pentasodium No concurrent radiotherapy Surgery: See Disease Characteristics At least 4 weeks since prior major surgery and recovered No concurrent surgery Other: No other concurrent anticancer treatment At least 28 days since investigational drugs, including analgesics or antiemetics No other investigational drugs during and for 28 days after study No concurrent drugs that induce or inhibit CYP3A enzyme No concurrent herbal preparations (e.g., PC-SPES)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-06; Primary Completion 2001-08 (Actual); Study Completion 2001-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L. DeJager, MD, FACP, Study Chair — Daiichi Sankyo
Locations (2):
- United States (2):
  - U.S. Oncology Research Inc., Houston, Texas
  - Institute for Drug Development, San Antonio, Texas